CLINICAL TRIAL: NCT01510912
Title: A Multicenter, Open-Label, Safety Study of Diclofenac [Test] Capsules in Subjects With Osteoarthritis of the Knee or Hip
Brief Title: Open-Label Study of Diclofenac Capsules to Treat Osteoarthritis Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIC3-08-06
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diclofenac Capsules 35 mg bid or tid (Experimental)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — 35 mg bid or tid Capsules

SUMMARY:
The purpose of this study is to evaluate the safety of Diclofenac [Test] Capsules for the treatment of osteoarthritis pain of the knee or hip.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ [greater than or equal to] 40 years of age
* If a participant in the previous DIC3-08-05 study, completed the study and did not discontinue for lack of efficacy or safety
* Has a diagnosis of OA of the hip or knee with ongoing knee and/or articular hip pain
* Is a current chronic user of nonsteroidal anti-inflammatory drugs (NSAIDs) and/or acetaminophen for his/her OA pain and is anticipated to benefit from continuous treatment with therapeutic doses of NSAIDs. A current chronic user is defined as a subject who has used these treatments for ≥ [greater than or equal to] 20 days of the last 30 days before screening

Exclusion Criteria:

* Has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any nonsteroid anti-inflammatory drugs (NSAIDs), including diclofenac
* Requires chronic use of opioid or opioid combination products to control OA pain of the knee or hip
* Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease
* Has significant difficulties swallowing capsules or is unable to tolerate oral medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Agaiby, MD, Principal Investigator — Clinical Investigation Specialists, Inc; Eddie Armas, MD, Principal Investigator — Well Pharma Medical Medical Research, Corporation; Matthew Barton, MD, Principal Investigator — Office of Matthew Barton, MD; David Bouda, MD, Principal Investigator — Heartland Clinical Research; Venkata Challa, MD, Principal Investigator — Peters Medical Research; John Champlin, MD, Principal Investigator — Med Center; Francisco Chevres, MD, Principal Investigator — Pinnacle Trials, Inc; Melanie Christina, MD, Principal Investigator — Clinical Investigations of Texas, LLC; James R Clark, MD, Principal Investigator — Charlottesville Medical Research Center, LLC; Stephen Daniels, DO, Principal Investigator — Premier Research Group - Austin; Richard R Eckert, MD, Principal Investigator — Hypothetest, LLC; Brandon Essink, MD, Principal Investigator — Meridian Clinical Research; Richard M Glover, MD, Principal Investigator — Heartland Research Associates, LLC; Kent S Hoffman, DO, Principal Investigator — Alliance Clinical Research; Curtis S Horn, MD, Principal Investigator — Quality Research Inc; Raymond E Jackson, MD, Principal Investigator — Quest Research Institute; Jeffry Jacqmein, MD, Principal Investigator — Jacksonville Center For Clinical Research; Enrico Jones, MD, Principal Investigator — Triad Clinical Research; Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research; Kevin Kuettel, MD, Principal Investigator — Acri-Phase I, LLC; Gregory F Lakin, DO, Principal Investigator — Professional Research Network of Kansas, LLC; Theresia Lee, MD, Principal Investigator — Progressive Clinical Research; Sathish Modugu, MD, Principal Investigator — Drug Trials America; Julie A Mullen, DO, Principal Investigator — Sterling Research Group, Ltd; Kashyap Patel, MD, Principal Investigator — Peninsula Research, Inc; Kyle Patrick, DO, Principal Investigator — Premier Research Group - Phoenix; Antoinette A Pragalos, MD, Principal Investigator — Community Research; Larry D Reed, MD, Principal Investigator — Healthcare Research; Eli M Roth, MD, Principal Investigator — Sterling Research Group, Ltd; Douglas R Schumacher, MD, Principal Investigator — Radiant Research, Inc; Mark Stich, DO, Principal Investigator — Westside Center for Clinical Research; Bradley Swenson, MD, Principal Investigator — Radiant Research, Inc; Gary Tarshis, MD, Principal Investigator — Expresscare Clinical Research; Haydn M Thomas, MD, Principal Investigator — Clinical Trials Technology Inc; Cindy Tuten, MD, Principal Investigator — Clinical Study Center of Asheville, LLC; Larkin T Wadsworth, MD, Principal Investigator — Sundance Clinical Research, LLC; Robert J Wagner, MD, Principal Investigator — Community Research; Larry S Watkins, MD, Principal Investigator — Lynn Institute of the Ozarks; Tamela Zimmerman, MD, Principal Investigator — Community Research; Marvin Tark, MD, Principal Investigator — Drug Studies America
Locations (38):
- United States (38):
  - Premier Research Group - Phoenix, Phoenix, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Acri-Phase I, LLC, Anaheim, California
  - Med Center, Carmichael, California
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Well Pharma Medical Research, Corporation, Miami, Florida
  - Peninsula Research, Inc, Ormond Beach, Florida
  - Alliance Clinical Research, Winter Park, Florida
  - Pinnacle Trials, Inc, Atlanta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Heartland Research Associates, LLC, Newton, Kansas
  - Clinical Trials Technology Inc, Prairie Village, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Quest Research Institute, Bingham Farms, Michigan
  - Healthcare Research, Florissant, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Office of Matthew Barton, MD, Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Triad Clinical Research, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Radiant Research, Inc, Columbus, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Radiant Research, Inc, Anderson, South Carolina
  - Premier Research Group - Austin, Austin, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Hypothetest, LLC, Roanoke, Virginia

REFERENCES:
- [Derived] Altman RD, Strand V, Hochberg MC, Gibofsky A, Markenson JA, Hopkins WE, Cryer B, Kivitz A, Nezzer J, Imasogie O, Young CL. Low-dose SoluMatrix diclofenac in the treatment of osteoarthritis: A 1-year, open-label, Phase III safety study. Postgrad Med. 2015 Jun;127(5):517-28. doi: 10.1080/00325481.2015.1040716. Epub 2015 Apr 27. PMID 25913498

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac 35 mg Capsules: Participants were administered Diclofenac 35 mg capsules two times daily and could either be uptitrated to three times daily or remain at two times daily. Participants who were uptitrated to three times daily were allowed to downtitrate to two times daily either temporarily or permanently. Participants could change regimens between two and three times daily as often as needed, with the approval of the investigator.
Period: Overall Study
Arm/Group | Diclofenac 35 mg Capsules
Started | 602
Completed | 360
Not Completed | 242
Not completed — Adverse Event | 99
Not completed — Lack of Efficacy | 12
Not completed — Non-compliance with trial drug | 23
Not completed — Withdrawal by Subject | 49
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 27
Not completed — Lost to Follow-up | 26
Not completed — Other, including joint replacement | 5

BASELINE CHARACTERISTICS:
Population: The safety population included all subjects who were treated with at least 1 dose of trial drug. Of the 602 subjects who started the study, 601 received at least 1 dose of trial drug.
Arm/Group | Diclofenac 35 mg Capsules
Number analyzed (Participants) | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 372
  Male | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 561
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race; therefore, some subjects are counted multiple times.
  participants
    American Indian or Alaska Native | 2
    Asian | 6
    Black or African American | 89
    White | 506
    Other | 1
Weight [Mean (Standard Deviation); unit: kg] | 87.93 (17.005)
Height [Mean (Standard Deviation); unit: cm] | 169.25 (9.898)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.574 (4.9818)
Baseline Mental Component Score of the Short Form-36 Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Short Form-36 is a validated 11-item health survey that assesses subject views about his/her functional health and well-being. The survey consists of 36 questions concerning daily or recent health-related activities and assesses 8 health domains using scaled scores. The mental component score is composed of a subset of the 8 health domains. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability.
  units on a scale | 52.0 (9.60)
Baseline Physical Component Score of the Short Form-36 Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Short Form-36 is a validated 11-item health survey that assesses subject views about his/her functional health and well-being. The survey consists of 36 questions concerning daily or recent health-related activities and assesses 8 health domains using scaled scores. The physical component score is composed of a subset of the 8 health domains. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability.
  units on a scale | 39.5 (7.72)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Diclofenac 35 mg Capsules as Assessed by the Incidence of Adverse Events From Baseline to Week 52 or Early Termination
Description: The safety of Diclofenac 35 mg capsules was assessed by the number of subjects with treatment-emergent adverse events (TEAEs), severe TEAEs, and serious adverse events.
Time Frame: Baseline to Week 52/Early Termination
Measure: Number; unit: participants
Arm/Group | Diclofenac 35 mg Capsules
Number analyzed (Participants) | 601
participants
  Subjects with at least 1 TEAE | 451
  Subjects with at least 1 severe TEAE | 41
  Subjects with at least 1 serious adverse event | 42

2. Other Pre Specified Outcome: Mean Short Form-36 Physical Component Summary Scores at Week 52/Early Termination (ET) and Change From Baseline to Week 52/ET
Description: The Short Form-36 is a validated 11-item health survey that assesses subject views about his/her functional health and well-being. The survey consists of 36 questions concerning daily or recent health-related activities and assesses 8 health domains using scaled scores. The physical component score is composed of a subset of the 8 health domains. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability.
Time Frame: Baseline to Week 52/Early Termination
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac 35 mg Capsules
Number analyzed (Participants) | 555
units on a scale
  Mean score at Week 52/early termination (ET) | 44.2 (8.29)
  Mean change from baseline to Week 52/ET | 4.5 (6.89)

3. Other Pre Specified Outcome: Mean Short Form-36 Mental Component Summary Scores at Week 52/Early Termination (ET) and Change From Baseline to Week 52/ET
Description: The Short Form-36 is a validated 11-item health survey that assesses subject views about his/her functional health and well-being. The survey consists of 36 questions concerning daily or recent health-related activities and assesses 8 health domains using scaled scores. The mental component score is composed of a subset of the 8 health domains. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability.
Time Frame: Baseline to Week 52/Early Termination
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac 35 mg Capsules
Number analyzed (Participants) | 555
units on a scale
  Mean score at Week 52/early termination (ET) | 52.3 (9.44)
  Change from baseline to Week 52/ET | 0.1 (8.41)

ADVERSE EVENTS:
Arm/Group | Diclofenac 35 mg Capsules
Serious Adverse Events (participants affected / at risk) | 42/601
Other Adverse Events (participants affected / at risk) | 191/601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac 35 mg Capsules (N=601)
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Hyperparathyroidism (Endocrine disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Intestinal strangulation (Gastrointestinal disorders) | 1
Pancreatitis (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 2
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dural tear (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Finger amputation (Surgical and medical procedures) | 1
Carotid artery stenosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac 35 mg Capsules (N=601)
Upper respiratory tract infection (Infections and infestations) | 47
Headache (Nervous system disorders) | 46
Urinary tract infection (Infections and infestations) | 44
Diarrhea (Gastrointestinal disorders) | 37
Nasopharyngitis (Infections and infestations) | 34
Nausea (Gastrointestinal disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No